CLINICAL TRIAL: NCT06722222
Title: A New Surgical Method for Treating Tandem Carotid Lesions: Gao's Triple Eversion Carotid Endarterectomy
Brief Title: Gao's Triple Eversion Carotid Endarterectomy
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1043
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenosis; tandem carotid lesion
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- tandem carotid lesions: Extracranial tandem carotid lesions (TCLs) refer to two or more severe stenoses/occlusions in two or more locations in the carotid artery. TCLs are indicated for surgical intervention but are difficult to resolve by conventional carotid endarterectomy
  Interventions: Procedure: Gao's triple eversion carotid endarterectomy

INTERVENTIONS:
Procedure: Gao's triple eversion carotid endarterectomy — The carotid sheath is dissected in front of the sternocleidomastoid muscle to expose sufficient lengths of the CCA, ECA, and ICA. After raising the systolic blood pressure to 180 mmHg and intravenously injecting 1 mg/kg heparin, the superior thyroid artery is lapped and severed, and the CCA is occluded proximally to the CCA plaque, based on the plaque location shown by preoperative CTA and by intraoperative arterial exploration. Subsequently, the ECA and ICA are blocked individually. The ICA is cut diagonally at the CCA fork and the ECA is transected approximately 5 mm above its beginning. The plaque is removed with tweezers after eversion of the ICA. This process is repeated for the ECA. Finally, the long segment of plaque in the CCA is stripped proximally, followed by thorough removal of the debris on the peeling surface using heparin irrigation.

SUMMARY:
Carotid endarterectomy (CEA), an important surgical approach for managing carotid plaque, has evolved over more than 70 years but still cannot be applied to all tandem carotid lesions (TCLs) because of the wide range of these lesions. Herein, the investigators introduce an innovative CEA, Gao's triple eversion CEA (GTE-CEA), for the treatment of TCLs.

DETAILED DESCRIPTION:
The investigators retrospectively reviewed the charts of patients who underwent GTE-CEA performed by the same group of vascular surgeons since 17 September, 2021. Patients who did not meet the diagnostic criteria for carotid artery stenosis (CAS); those with asymptomatic CAS < 50%, preoperatively confirmed by digital subtraction angiography (DSA) or computed tomography angiography (CTA); and those with stenosis at the opening of the common carotid artery (CCA) were excluded from our study.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for TCL stenosis.
* Above 70% asymptomatic CCA and ICA stenosis or > 50% symptomatic CAS confirmed by DSA or CTA before surgery

Exclusion Criteria:

* Did not meet the diagnostic criteria for CAS
* Asymptomatic CAS < 50% (as confirmed by DSA or CTA before surgery)
* With stenosis at the opening of the CCA.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extracranial tandem carotid lesions (TCLs) refer to two or more severe stenoses/occlusions in two or more locations in the carotid artery. TCLs are indicated for surgical intervention but are difficult to resolve by conventional carotid endarterectomy (CEA). The incidence of stenosis in the common carotid artery (CCA) combined with that in the internal carotid artery (ICA) reportedly accounts for approximately 5% of all CAS cases.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2031-09-20 (Estimated); Study Completion 2031-09-20 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Until the end of the study, an average of 3 years
  Digital subtraction angiography (DSA) or computed tomography angiography showed carotid artery recanalization and no risk complications such as stroke

CONTACTS AND LOCATIONS:
Overall Officials: Zhiwei Gao, Dr., Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators are preparing their submission and they will share it in the receiving magazine.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will become available after the submission is received by a magezine.
Access Criteria: The data that support the findings of this study are available from Zhiwei Gao upon reasonable request.

REFERENCES:
- [Background] Georg Y, Psathas E, Alomran F, Gaudric J, Chiche L, Koskas F. Double eversion carotid endarterectomy of tandem carotid lesions. Ann Vasc Surg. 2014 Jul;28(5):1186-91. doi: 10.1016/j.avsg.2013.07.018. Epub 2013 Oct 27. PMID 24495326
- [Background] Davidovic LB, Tomic IZ. Eversion Carotid Endarterectomy : A Short Review. J Korean Neurosurg Soc. 2020 May;63(3):373-379. doi: 10.3340/jkns.2019.0201. Epub 2020 Mar 2. PMID 32114754
- [Background] Marko M, Cimflova P, Poppe AY, Kashani N, Singh N, Ospel J, Mayank A, van Adel B, McTaggart RA, Nogueira RG, Demchuk AM, Rempel JL, Joshi M, Zerna C, Menon BK, Tymianski M, Hill MD, Goyal M, Almekhlafi MA; ESCAPE-NA1 investigators. Management and outcome of patients with acute ischemic stroke and tandem carotid occlusion in the ESCAPE-NA1 trial. J Neurointerv Surg. 2022 May;14(5):neurintsurg-2021-017474. doi: 10.1136/neurintsurg-2021-017474. Epub 2021 May 4. PMID 33947770
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Assis Z, Menon BK, Goyal M, Demchuk AM, Shankar J, Rempel JL, Roy D, Poppe AY, Yang V, Lum C, Dowlatshahi D, Thornton J, Choe H, Burns PA, Frei DF, Baxter BW, Hill MD; ESCAPE Trialists. Acute ischemic stroke with tandem lesions: technical endovascular management and clinical outcomes from the ESCAPE trial. J Neurointerv Surg. 2018 May;10(5):429-433. doi: 10.1136/neurintsurg-2017-013316. Epub 2017 Oct 11. PMID 29021311
- [Background] Anadani M, Spiotta AM, Alawieh A, Turjman F, Piotin M, Haussen DC, Nogueira RG, Papanagiotou P, Siddiqui AH, Lapergue B, Dorn F, Cognard C, Ribo M, Psychogios MN, Labeyrie MA, Mazighi M, Biondi A, Anxionnat R, Bracard S, Richard S, Gory B; TITAN (Thrombectomy In TANdem Lesions) Investigators. Emergent Carotid Stenting Plus Thrombectomy After Thrombolysis in Tandem Strokes: Analysis of the TITAN Registry. Stroke. 2019 Aug;50(8):2250-2252. doi: 10.1161/STROKEAHA.118.024733. Epub 2019 Jun 17. PMID 31577899
- [Background] DeCarlo C, Tanious A, Boitano LT, Mohebali J, Stone DH, Clouse WD, Conrad MF. Simultaneous treatment of common carotid lesions increases the risk of stroke and death after carotid artery stenting. J Vasc Surg. 2021 Aug;74(2):592-598.e1. doi: 10.1016/j.jvs.2020.12.089. Epub 2021 Feb 2. PMID 33545307
- [Background] Rouleau PA, Huston J 3rd, Gilbertson J, Brown RD Jr, Meyer FB, Bower TC. Carotid artery tandem lesions: frequency of angiographic detection and consequences for endarterectomy. AJNR Am J Neuroradiol. 1999 Apr;20(4):621-5. PMID 10319972
- [Background] CRAWFORD ES, DEBAKEY M, FIELDS WS, MORRIS GC Jr, COOLEY DA. Surgical considerations in the treatment of cerebral arterial insufficiency; scientific exhibit. Postgrad Med. 1959 Aug;26(2):227-37. doi: 10.1080/00325481.1959.11712569. No abstract available. PMID 13675020